CLINICAL TRIAL: NCT06756633
Title: Evaluation of Respiratory Functions, Thoracoabdominal Movements, and Exercise Capacity in Neuromuscular Diseases
Brief Title: Respiratory Functions, Thoracoabdominal Movements and Exercise Capacity in Neuromuscular Diseases
Status: Recruiting | Type: Observational
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Bilge Taskin Gurel, Principal Investigator, Lokman Hekim University
Other Study IDs: LokmanHekimUniv
Record Dates: First submitted 2024-05-28; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Neuromuscular Diseases in Children; Respiratory Function Impaired; Respiratory Insufficiency; Duchenne Muscular Dystrophy; Spinal Muscular Atrophy; Plethysmography
Keywords: Duchenne muscular dystrophy; Spinal muscular atrophy; respiratory function tests; plethysmography
MeSH Terms: conditions — Respiratory Insufficiency; Muscular Dystrophy, Duchenne; Muscular Atrophy, Spinal | interventions — Respiratory Physiological Phenomena; Hand Strength

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Duchenne muscular dystrophy: Participants in this group will be clinically diagnosed with Duchenne Muscular Dystrophy. Eligibility criteria include being over 5 years of age, having the ability to breathe independently without mechanical support, and voluntarily agreeing to participate in the study. Participants will be excluded if they have cognitive problems that may affect test results, have undergone pulmonary surgery, or have advanced heart failure.
  Interventions: Other: Respiratory Function Test; Other: Structured light plethysmography; Other: 6 Minute Walking Test; Other: 6-Minute Peg Board Ring Test; Other: Hand Grip Strength
- Spinal muscular atrophy: This group will include participants with a clinical diagnosis of Spinal Muscular Atrophy. Similar to the DMD group, eligibility criteria include being over 5 years old, having independent respiratory function, and providing informed consent for study participation. Exclusion criteria for this group are the presence of cognitive impairments that could influence evaluation results, a history of pulmonary surgery, or advanced heart failure.
  Interventions: Other: Respiratory Function Test; Other: Structured light plethysmography; Other: 6 Minute Walking Test; Other: 6-Minute Peg Board Ring Test; Other: Hand Grip Strength
- Healthy controls: The control group will consist of healthy participants over 5 years of age with no known neuromuscular or respiratory conditions. Participants must be capable of independent breathing and willing to participate in the study. Individuals with cognitive impairments, a history of pulmonary surgery, or any underlying medical condition that could interfere with study outcomes will be excluded from this group.
  Interventions: Other: Respiratory Function Test; Other: Structured light plethysmography; Other: 6 Minute Walking Test; Other: 6-Minute Peg Board Ring Test; Other: Hand Grip Strength

INTERVENTIONS:
Other: Respiratory Function Test — A spirometer (microQuark, COSMED) will be used to assess respiratory functions. During a forced expiratory maneuver after a deep, full inspiration, airway and lung volumes are measured. During the measurement, a deep inspiration followed by a strong, fast, and continuous expiration until unable to exhale anymore should be performed. The expiration time should be at least 6 seconds, and if necessary, extended up to 15 seconds. More than eight repetitions at one time are not recommended.
Other: Structured light plethysmography — Participants' thoracoabdominal movements will be assessed using the PneumoCare device that measures with the SLP technique. The evaluation begins with positioning participants wearing a white tank top, t-shirt, or with a bare chest. In our study, measurements will be taken with participants seated, supported by their backs, and their chest area exposed. The participant's age, height, and weight information are entered into the system. After the participant is positioned, the lights of the SLP measuring device are set up 90-100 cm away to encompass the chest area. The light field, which is in a checkerboard pattern, rectangular or square, should align its upper edge with the participant's clavicles and its lower edge with the anterior-superior iliac spine. During this measurement, the participant is asked to look straight ahead and breathe normally for five minutes. At the end of the measurement, the three-dimensional movements of the chest and respiratory parameters are recorded.
Other: 6 Minute Walking Test — For Ambulatory Participants:
  Exercise capacity will be assessed using the Six-Minute Walk Test (6MWT). The test will be performed according to ATS/ERS guidelines . The test involves walking for six minutes at a submaximal level in a 20-meter corridor. Blood pressure, heart rate, respiratory rate, oxygen saturation, and dyspnea, general fatigue, and leg fatigue according to the Modified BORG Scale (MBS) will be assessed before and after the test. Participants can stop and rest during the test. In such cases, the test duration is paused, and the rest time is recorded, then the test resumes from where it was left off. The distance walked in meters at the end of the test is recorded.
Other: 6-Minute Peg Board Ring Test — For Non-Ambulatory Participants:
  The 6-Minute Pegboard Ring Test will be used to assess upper extremity exercise capacity . Pre- and post-test evaluations of heart rate, blood pressure, respiratory rate, and MBS for dyspnea and fatigue will be made. The board used for the test has a total of 6 holes spaced 10 cm apart horizontally and another set of 6 holes 20 cm below aligned with the top row. There are four 20 cm long iron rods suitable for the holes. A total of 20 rings suitable for the iron rods will be used. The iron rods will be placed in the designated holes according to the patients' shoulder width. An adjustable chair will be used to suit the patients' heights, and the distance between the chair and the board will be adjusted according to arm length. Patients will be asked to place the rings from top to bottom and bottom to top with both hands simultaneously. The total number of rings placed in six minutes will be recorded in units.
Other: Hand Grip Strength — Hand grip strength will be measured using a digital hand dynamometer (CAMRY Digital Hand Dynamometer) . The device handle will be adjusted according to the participants' hand size. The test is conducted while seated, with the dominant upper extremity in 90 degrees of elbow flexion. Participants are asked to squeeze the dynamometer as strongly as possible. The value displayed on the dynamometer is recorded. The measurement is repeated three times, and the average of the three measurements is taken to determine the participant's hand grip strength. The measurement takes five minutes and does not need to be repeated.

SUMMARY:
The clinical trial titled "Investigation of Respiratory Functions, Thoracoabdominal Movements, and Exercise Capacity in Neuromuscular Diseases" aims to evaluate the respiratory functions, thoracoabdominal movements, and exercise capacity in children with Duchenne Muscular Dystrophy (DMD) and Spinal Muscular Atrophy (SMA) compared to healthy controls. The study will use spirometry, structured light plethysmography (SLP), the six-minute walk test, and the six-minute pegboard ring test to assess these functions. This trial will be conducted at the Lokman Hekim University Muscle and Nerve Diseases Application and Research Center from May 2024 to Dec 2025.

DETAILED DESCRIPTION:
This cross-sectional study will be conducted at the Lokman Hekim University Muscle and Nerve Diseases Application and Research Center over a 20-month period from May 2024 to December 2025. The study will include a total of 42 children, with three groups of 14 participants each: children diagnosed with Duchenne Muscular Dystrophy (DMD), children diagnosed with Spinal Muscular Atrophy (SMA), and a healthy control group. The study is designed to evaluate key respiratory, functional, and muscular parameters in these groups.

Respiratory parameters will be assessed using spirometry and Structured Light Plethysmography (SLP). Spirometry will involve maximal inspiratory and expiratory maneuvers to measure lung volumes and capacities, conducted under standardized conditions and monitored by a trained technician. SLP will be conducted using the PneumoCare device, a non-invasive system that measures thoracoabdominal movement during tidal breathing. A grid of light will be projected onto the chest to capture three-dimensional movement patterns over a five-minute period with participants in a seated position.

Functional and muscular assessments will include the Six-Minute Walk Test (6MWT), the Six-Peg Board Ring Test (6PBRT), and hand grip strength measurements. The 6MWT will be conducted in a 20-meter corridor, where participants will walk for six minutes at their own pace, with heart rate, blood pressure, and oxygen saturation recorded before and after the test. The 6PBRT will assess upper-limb endurance and strength through the timed movement of rings across a pegboard, with accuracy and task duration recorded. Hand grip strength will be measured using a handheld dynamometer, with participants performing three trials, and the highest value noted for analysis.

Data analysis will be performed using IBM SPSS Statistics version 23.0. Descriptive statistics will summarize the demographic and clinical characteristics of participants. Group comparisons will be conducted using independent samples t-tests, Mann-Whitney U tests for non-normally distributed variables, and one-way ANOVA for multi-group comparisons. Correlations between variables will be assessed using Pearson or Spearman correlation coefficients, depending on the distribution of the data. A significance threshold of p<0.05 will be applied, with Bonferroni corrections for multiple comparisons as needed.

Ethical approval for this study was granted by the Lokman Hekim University Scientific Research Ethics Committee (approval number: 2024114). All participants and their legal guardians will provide informed consent prior to enrollment, and all data will be anonymized and securely stored in compliance with the General Data Protection Regulation (GDPR). The study will follow Good Clinical Practices (GCP) and adhere to the ethical principles of the Declaration of Helsinki.

The primary objective is to evaluate and compare respiratory, functional, and muscular parameters in children with DMD and SMA against those in healthy peers. The study aims to identify distinctive patterns and impairments within the patient groups, which could provide insights for developing targeted therapeutic interventions.

ELIGIBILITY:
1. Duchenne Muscular Dystrophy (DMD)

   -Inclusion Criteria: Clinically diagnosed with Duchenne Muscular Dystrophy. Age above 5 years. Able to breathe independently. Willing to participate in the study.

   -Exclusion Criteria: Presence of cognitive problems that affect the assessment results. History of pulmonary surgery. Advanced heart failure.
2. Spinal Muscular Atrophy (SMA)

   -Inclusion Criteria: Clinically diagnosed with Spinal Muscular Atrophy. Age above 5 years. Able to breathe independently. Willing to participate in the study.

   -Exclusion Criteria: Presence of cognitive problems that affect the assessment results. History of pulmonary surgery. Advanced heart failure.
3. Healthy Controls

   * Inclusion Criteria:

No diagnosis of neuromuscular diseases. Age above 5 years. Able to breathe independently. Willing to participate in the study.

-Exclusion Criteria: Presence of cognitive problems that affect the assessment results. History of pulmonary surgery. Advanced heart failure.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study involves three groups: children with Duchenne Muscular Dystrophy (DMD), children with Spinal Muscular Atrophy (SMA), and healthy controls.
  Group 1: This group includes children clinically diagnosed with DMD, a progressive neuromuscular disorder caused by dystrophin gene mutations. Participants are over 5 years old and can breathe independently, including both ambulatory and non-ambulatory children.
  Group 2:This group comprises children diagnosed with SMA, a genetic disorder leading to motor neuron degeneration. Participants are over 5 years old and can breathe independently, and non-ambulatory children.
  Group 3: The control group consists of healthy children over 5 years old with no neuromuscular diseases. Their inclusion allows for comparative analysis.
  The study aims to enroll 42 participants, with 14 in each group, ensuring 80% study power with a 5% Type 1 error rate.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | Baseline (Day 1)
  Forced Vital Capacity (FVC) measures the maximum volume of air that a participant can exhale forcefully after taking a deep breath. This measure reflects lung capacity.
Forced Expiratory Volume in 1 Second (FEV1) | Baseline (Day 1)
  Forced Expiratory Volume in 1 second (FEV1) represents the volume of air that can be forcefully exhaled in one second. This measure evaluates airway function and obstruction.
Peak Expiratory Flow (PEF) | Baseline (Day 1)
  Peak Expiratory Flow (PEF) assesses the maximum speed of air expelled during expiration, indicating airway resistance.
FEV1/FVC Ratio | Baseline (Day 1)
  The ratio of FEV1 to FVC, expressed as a percentage, evaluates airflow limitation severity.
6-Minute Walk Test (6MWT) | Baseline (Day 1)
  The 6-Minute Walk Test (6MWT) assesses lower-limb functional capacity by measuring the total distance a participant can walk in six minutes at their own pace on a flat, 20-meter corridor. The test evaluates endurance and physical capacity. Heart rate, blood pressure, and oxygen saturation will be measured immediately before and after the test to assess physiological responses.
Thoracoabdominal movement | 8 min
  Detection of thoracoabdominal asyncrony and analysis of the kinematics of breathing
Hand Grip Strength | 5 min
  Digital hand dynamometer
6-Minute Peg Board Ring Test (6PBRT) | Baseline (Day 1)
  The 6-Minute Peg Board Ring Test (6PBRT) evaluates upper-limb endurance and strength. Participants will move rings between pegs on a pegboard for six minutes, with the total number of rings successfully placed recorded as the outcome. This test is designed to assess upper-limb functional capacity and fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The IPD collected in this study is securely stored in the Lokman Hekim University database. Participants' demographic information and the study's measurement results can be shared by the responsible investigator upon receipt of a valid request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting information will be available starting 6 months after the study's completion date and will remain accessible for 5 years.
Access Criteria: Access to IPD and supporting information will be granted to researchers with a valid scientific purpose, subject to approval by the responsible investigator. Requests must include a detailed research proposal outlining the objectives and intended use of the data. Approved researchers will be provided access to anonymized data through a secure data-sharing platform.